CLINICAL TRIAL: NCT06559085
Title: Posterior Versus Lateral Laparoscopic Mesh Rectopexy for the Management of Complete Rectal Prolapse
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Mohamed Ahmed Mohamed Makhlouf, Assistant Lecturer of General Surgery, Assiut University, Assiut, Egypt, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-2024-100197
Record Dates: First submitted 2024-08-10; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Posterior Laparoscopic; Lateral Laparoscopic; Rectopexy; Complete Rectal Prolapse
MeSH Terms: interventions — Water Wells

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laproscopic posterior mesh rectopexy (Wells or LPMR) (Experimental): After complete rectal mobilization, a mesh is inserted between the sacrum and the posterior rectum, sutured into the rectum, and fixed to the promontory. The mortality rates ranged from 0% to 1.2%, and recurrence rates ranged from 0% to 11% There was an overall improvement in continence (74%-100%), with conflicting results regarding constipation. New-onset constipation in 5% to 44% of patients was reported
  Interventions: Procedure: Laproscopic posterior mesh rectopexy (Wells or LPMR)
- Laparoscopic lateral mesh rectopexy (Orr-Loygue) (Experimental): This procedure involves complete mobilization of the rectum with two mesh strips sutured laterally to the rectal wall on both sides, and they were suspended to the promontory. There are several studies on this procedure using a laparoscopic approach. Lechaux et al. performed laparoscopic Orr-Loygue rectopexy in 35 patients. Incontinence improved in 27% of patients, and constipation improved in 19% but worsened in 27%. The recurrence rate was 3% (1/35) after a mean follow-up of 36 months. A study on 46 patients with laparoscopic Orr-Loygue procedure with posterior mobilization found a significant reduction in incontinence score after 1 year, but there were no changes in the use of laxatives. The recurrence rate was 4% after a median follow-up of 1.5 years.
  Interventions: Procedure: Laparoscopic lateral mesh rectopexy (Orr-Loygue)

INTERVENTIONS:
Procedure: Laproscopic posterior mesh rectopexy (Wells or LPMR) — After complete rectal mobilization, a mesh is inserted between the sacrum and the posterior rectum, sutured into the rectum, and fixed to the promontory. The mortality rates ranged from 0% to 1.2%, and recurrence rates ranged from 0% to 11% There was an overall improvement in continence (74%-100%), with conflicting results regarding constipation. New-onset constipation in 5% to 44% of patients was reported
  Arms: Laproscopic posterior mesh rectopexy (Wells or LPMR)
Procedure: Laparoscopic lateral mesh rectopexy (Orr-Loygue) — This procedure involves complete mobilization of the rectum with two mesh strips sutured laterally to the rectal wall on both sides, and they were suspended to the promontory. There are several studies on this procedure using a laparoscopic approach. Lechaux et al. performed laparoscopic Orr-Loygue rectopexy in 35 patients. Incontinence improved in 27% of patients, and constipation improved in 19% but worsened in 27%. The recurrence rate was 3% (1/35) after a mean follow-up of 36 months. A study on 46 patients with laparoscopic Orr-Loygue procedure with posterior mobilization found a significant reduction in incontinence score after 1 year, but there were no changes in the use of laxatives. The recurrence rate was 4% after a median follow-up of 1.5 years
  Arms: Laparoscopic lateral mesh rectopexy (Orr-Loygue)

SUMMARY:
Aim of the study is to evaluate the outcomes of two different methods of mesh placement during laparoscopic rectopexy for the management of complete rectal prolapse lateral versus posterior mesh rectopexy

DETAILED DESCRIPTION:
Rectal prolapse is the full-thickness prolapse of the rectum, in which the rectum passes externally beyond the anal sphincters. It is a somewhat rare condition, estimated to occur in less than 0.5% of the population. Rectal prolapse has a 9:1 female predominance, and while it is occasionally seen in younger individuals, the incidence increases with age.

Surgical approaches for rectal prolapse can be divided into perineal and abdominal approaches. Traditionally, a perineal procedure such as Delorme or Altemeir operation was commonly used in elderly or frail patients while an abdominal procedure such as rectopexy with or without resection was reserved for younger and fitter patients. The frequency of laparoscopic abdominal repair of rectal prolapse has increased in recent years, with mesh rectopexy being the most popular procedure.

The mesh rectopexy operation was first described by Ripstein10 in 1952. Again, after mobilization of the rectum, an anterior sling of synthetic material (either absorbable or non-absorbable) is placed in front of the rectum and sutured to the sacral promontory. The rationale for this is to restore the natural curve of the rectum, which reduces the effect of downward abdominal pressure. The use of a non-elastic synthetic graft provides a firm anterior fascial support even in patients with significant pelvic floor descent, returning the rectum to a normal anatomical position.

The act of mobilization, suture, and fibrosis keeps the rectum fixed in position as adhesions form, attaching the rectum to the presacral fascia. Although SR is considered a good option for the cure of rectal prolapse/IS in both men and women, some reviews of this procedure noted a better overall clinical outcome in men. This may be due to occult sphincter defects in women, and failure to detect these defects before surgery owing to the lack of routine endoanal ultrasonography in the earlier years of prolapse surgery

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 70 years.
* Both sexes.
* Patients with complete rectal prolapse.

Exclusion Criteria:

* Unfit for surgery
* Impaired coagulation profile
* Contraindication of laparoscopy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Operative time | Until the conclusion of the surgical procedure
  Operative time will be measured (Time Frame: from inflation of abdomen till deflation in laparoscopic repair and from skin incision up to skin closure in open repair)
Intraoperative injuries | Until the conclusion of the surgical procedure
  Intra operative injuries will be recorded including bowel or vascular injuries

SECONDARY OUTCOMES:
Improving of symptoms | 28 days after surgery
  Laparoscopic lateral mesh rectopexy versus posterior mesh rectopexy regarding to improving of symptoms will be recorded
Recurrence rate | 28 days after surgery
  Laparoscopic lateral mesh rectopexy versus posterior mesh rectopexy regarding to recurrence rate will be recorded The recurrence rate was 3% (1/35) after a mean follow-up of 36 months in laparoscopic lateral mesh rectopexy (Orr-Loygue) and recurrence rates ranged from 0% to 11% in laproscopic posterior mesh rectopexy (Wells or LPMR)
Complications | 28 days after surgery
  Complications will be recorded such as early as bleeding, incontinence, intestinal obstruction, late as constipation, sexual dysfunction, intestinal obstruction, erosion of mesh

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: ِِِAfter the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author